CLINICAL TRIAL: NCT04944901
Title: Randomized, Double-blind, Placebo-controlled, 28-Day Daily-dose Crossover Study of the Safety and Tolerability of SB-121 (Lactobacillus Reuteri With Sephadex® and Maltose) in Subjects, Ages 15 to 45 Years, Diagnosed With Autistic Disorder
Brief Title: 28-Day Daily-dose Crossover Study of the Safety and Tolerability of SB-121 (Lactobacillus Reuteri With Sephadex® and Maltose) in Subjects, Ages 15 to 45 Years, Diagnosed With Autistic Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scioto Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SBI-SB121-20-01
Record Dates: First submitted 2021-06-21; First posted 2021-06-30 (Actual); Results first posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-09

CONDITIONS: Autistic Disorder
Keywords: Lactobacillus reuteri; autistic disorder; microbiome
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SB-121 (Experimental): One dose of SB-121 daily for 28 days according to the treatment group to which they are allocated.
  Administration: Oral
  Interventions: Drug: SB-121
- Placebo (Placebo Comparator): One dose of placebo daily for 28 days according to the treatment group to which they are allocated.
  Administration: Oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SB-121 — SB-121 is a formulation of L. reuteri
  Arms: SB-121
Drug: Placebo — Placebo oral formulation
  Arms: Placebo

SUMMARY:
SB-121 is being developed for use in the treatment of autistic disorder (AD).

This study is a multiple-dose, randomized, double-blind, placebo-controlled, cross-over single-site Phase I study.

The primary objective is to evaluate the safety and tolerability of multiple doses of SB-121 in subjects ages 15 to 45 years with AD.

Additionally, multiple measures of AD, as well as mechanistic biomarkers, will be assessed in order to inform later stage trials.

ELIGIBILITY:
Inclusion Criteria:

* Subject/parent (or authorized designee) has provided written informed consent for the study.
* Subject is ≥15 and ≤45 years of age at the time of enrollment.
* Diagnosis of autistic disorder (AD) as confirmed by the gold standard clinical interview using Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria and administration of the Autism Diagnostic Observation Schedule-2.
* Subject, if female and of childbearing potential, is not lactating or pregnant.
* Subject, if female, is either not of childbearing potential or is practicing an acceptable effective method of birth control.
* Subject is willing to comply with all study requirements (including the requirements for stool sampling and biobanking) and to return to the study facility for the follow-up evaluations, as required.

Exclusion Criteria:

* Subject has known allergy or significant adverse reaction to L reuteri, Sephadex®, maltose, or related compounds.
* Subject has previously had GI surgery, intestinal obstruction, Clostridium difficile infection or diverticulitis.
* Subject has travelled outside of the USA in the 30 days prior to screening.
* Subject has had a diarrheal illness in 30 days prior to screening.
* Subject currently has a fever or active/uncontrolled gastrointestinal (GI) symptoms (e.g., nausea, vomiting, diarrhea, constipation, abdominal distention, abdominal pain/cramps, flatulence) or has had these within 14 days prior to screening. If the GI symptoms are stable, in the opinion of the investigator, the subject can be enrolled.
* Subject has any immunological/autoimmune disorder including, but not limited to, systemic lupus erythematosis, rheumatoid arthritis, Sjögren's syndrome, inflammatory bowel disease, or immunoglobulin-deficiency disorder, that would increase the risk to the subject or interfere with the evaluation of SB-121.
* Subject has a documented history of human immunodeficiency virus (HIV), hepatitis B and/or hepatitis C
* Subject has implanted prosthetic devices including prosthetic heart valves.
* Subject has taken, or is taking, any of the following prohibited medications:

  1. A proton pump inhibitor within 2 weeks prior to screening
  2. Use of supplemental probiotics within 2 weeks prior to screening except for yogurt
  3. Current use of immunosuppressive medications, including corticosteroids
  4. Treatment with monoclonal antibodies within 4 weeks prior to screening
  5. Systemic antibiotics within 2 weeks prior to screening
* Subject has diabetes mellitus or is prediabetic.
* Subject has received any IP (or investigational device) within 30 days prior to screening.
* Subject has any of the following laboratory test results at Screening:

  1. An absolute neutrophil count of <1.5 × 10^9/L
  2. alanine aminotransferase or aspartate aminotransferase >1.5 × upper limit normal (ULN), total bilirubin >1.5 × ULN (subjects with known Gilbert's Syndrome can be included)
  3. serum creatinine >1.5 × ULN
  4. any other abnormal laboratory test that is clinically significant in the judgment of the investigator.
* Subject has an unstable medical condition or is otherwise considered unreliable or incapable, in the opinion of the investigator, of complying with the requirements of the protocol.
* Subject tests positive for drugs of abuse in a urine drug screen at screening.
* Subject has a history of alcohol abuse.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Erickson, MD, Principal Investigator — University of Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmitt LM, Smith EG, Pedapati EV, Horn PS, Will M, Lamy M, Barber L, Trebley J, Meyer K, Heiman M, West KHJ, Hughes P, Ahuja S, Erickson CA. Results of a phase Ib study of SB-121, an investigational probiotic formulation, a randomized controlled trial in participants with autism spectrum disorder. Sci Rep. 2023 Mar 30;13(1):5192. doi: 10.1038/s41598-023-30909-0. PMID 36997569

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 15 participants were randomized in this crossover study.
Groups:
- Group 1 (SB-121 - Placebo): Treatment Period 1: One oral dose of SB-121 daily for 28 days. Treatment Period 2: One oral dose of placebo daily for 28 days.
  SB-121: SB-121 is a formulation of L. reuteri
- Group 2 (Placebo - SB-121): Treatment Period 1: One dose of oral placebo daily for 28 days. Treatment Period 2: One oral dose of SB-121 daily for 28 days.
  SB-121: SB-121 is a formulation of L. reuteri
Period: Treatment Period 1
Arm/Group | Group 1 (SB-121 - Placebo) | Group 2 (Placebo - SB-121)
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | Group 1 (SB-121 - Placebo) | Group 2 (Placebo - SB-121)
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (SB-121 - Placebo) | Group 2 (Placebo - SB-121) | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.1 (1.46) | 19.9 (4.09) | 20.0 (3.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 8 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 7 | 14
  Black or African American | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15
Height [Mean (Standard Deviation); unit: centimeters] | 177.96 (6.904) | 178.54 (6.280) | 178.27 (6.343)
Weight [Mean (Standard Deviation); unit: kilograms] | 69.67 (9.725) | 98.26 (40.006) | 84.92 (32.538)
Body mass index [Mean (Standard Deviation); unit: kilogram/meter squared] | 22.11 (3.859) | 31.29 (14.552) | 27.01 (11.606)
Autism Diagnostic Observation Schedule, 2nd edition (ADOS-2) Score [Mean (Standard Deviation); unit: ADOS-2 Score] — Scale = 0 to 28
  ADOS-2 is the gold-standard observation-based rating system used to aid assessment/diagnosis of autism. There are 5 different modules of the ADOS-2 that are used depending on the individual's age and language level (this study used modules 2, 3 and 4). For each Module there is a Total score and cut-off scores that indicate autism. Overall, a higher score = more behaviors associated with autism. However, cutoff scores differ depending on which module is used, as well as the individual's language level and/or age. All Modules range from a score of 0 to 28.
  ADOS-2 Score | 16.0 (4.40) | 13.6 (3.02) | 14.7 (3.79)
Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5 checklist) [Count of Participants; unit: Participants]
  Met criteria for Autism Spectrum Disorder | 7 | 8 | 15
  Not met criteria for Autism Spectrum Disorder | 0 | 0 | 0
Drug Abuse Screen via Urine [Count of Participants; unit: Participants]
  Negative | 6 | 6 | 12
  Positive | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Adverse Event of Special Interest (AESIs) and Adverse Events (AEs) Leading to Discontinuation
Description: Adverse event of special interest (AESIs) and adverse events (AEs) leading to discontinuation from the study are presented.
  Treatment Period 1: 2 participants reported 4 events in the SB-121 group and 3 participant reported 6 events in the placebo group.
  Treatment Period 2: 1 participant reported 3 events in the SB-121 group and 1 participant reported 4 events in the placebo group.
Time Frame: Approximately 98 days
Population: Safety Population
Measure: Number; unit: adverse events
Groups:
- SB-121: One dose of SB-121 daily for 28 days according to the treatment group to which they are allocated.
  Administration: Oral SB-121: SB-121 is a formulation of L. reuteri
- Placebo: One dose of placebo daily for 28 days according to the treatment group to which they are allocated.
  Administration: Oral Placebo: Placebo oral formulation
Arm/Group | SB-121 | Placebo
Number analyzed (Participants) | 15 | 15
adverse events
  Treatment Period 1 : Adverse events leading to discontinuation: number analyzed (Participants) | 7 | 8
  Treatment Period 1 : Adverse events leading to discontinuation | 0 | 0
  Treatment Period 1 : Diarrhoea (AESI): number analyzed (Participants) | 7 | 8
  Treatment Period 1 : Diarrhoea (AESI) | 1 | 2
  Treatment Period 1 : Abdominal pain (AESI): number analyzed (Participants) | 7 | 8
  Treatment Period 1 : Abdominal pain (AESI) | 0 | 2
  Treatment Period 1 : Abdominal pain upper (AESI): number analyzed (Participants) | 7 | 8
  Treatment Period 1 : Abdominal pain upper (AESI) | 2 | 0
  Treatment Period 1 : Nausea (AESI): number analyzed (Participants) | 7 | 8
  Treatment Period 1 : Nausea (AESI) | 1 | 0
  Treatment Period 1 : Vomiting (AESI): number analyzed (Participants) | 7 | 8
  Treatment Period 1 : Vomiting (AESI) | 0 | 2
  Treatment Period 2 : Adverse events leading to discontinuation: number analyzed (Participants) | 8 | 7
  Treatment Period 2 : Adverse events leading to discontinuation | 0 | 0
  Treatment Period 2 : Diarrhoea (AESI): number analyzed (Participants) | 8 | 7
  Treatment Period 2 : Diarrhoea (AESI) | 3 | 3
  Treatment Period 2 : Abdominal pain (AESI): number analyzed (Participants) | 8 | 7
  Treatment Period 2 : Abdominal pain (AESI) | 0 | 0
  Treatment Period 2 : Abdominal pain upper (AESI): number analyzed (Participants) | 8 | 7
  Treatment Period 2 : Abdominal pain upper (AESI) | 0 | 0
  Treatment Period 2 : Nausea (AESI): number analyzed (Participants) | 8 | 7
  Treatment Period 2 : Nausea (AESI) | 0 | 0
  Treatment Period 2 : Vomiting (AESI): number analyzed (Participants) | 8 | 7
  Treatment Period 2 : Vomiting (AESI) | 0 | 1

2. Primary Outcome: Sephadex Microspheres in the Stool
Description: The presence of Sephadex microspheres in the stool was assessed.
  The number of participants with data available at each stage are presented.
Time Frame: Period 1: Days 1 (pre-dose), 28 and 35; Period 2: Days 28 and 42 (period = 28 days and 14 days wash-out)
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | SB-121 | Placebo
Number analyzed (Participants) | 15 | 15
Participants
  Period 1 Day 1: number analyzed (Participants) | 3 | 3
  Period 1 Day 1: Sephadex Positive | 2 | 1
  Period 1 Day 1: Sephadex Negative | 1 | 2
  Period 1 Day 28: number analyzed (Participants) | 6 | 5
  Period 1 Day 28: Sephadex Positive | 6 | 5
  Period 1 Day 28: Sephadex Negative | 0 | 0
  Period 1 Day 35/Washout: number analyzed (Participants) | 3 | 4
  Period 1 Day 35/Washout: Sephadex Positive | 2 | 2
  Period 1 Day 35/Washout: Sephadex Negative | 1 | 2
  Period 2 Day 28/End of treatment: number analyzed (Participants) | 4 | 1
  Period 2 Day 28/End of treatment: Sephadex Positive | 4 | 1
  Period 2 Day 28/End of treatment: Sephadex Negative | 0 | 0
  Period 2 Day 42/Poststudy Washout: number analyzed (Participants) | 3 | 3
  Period 2 Day 42/Poststudy Washout: Sephadex Positive | 0 | 1
  Period 2 Day 42/Poststudy Washout: Sephadex Negative | 3 | 2

3. Primary Outcome: Symptomatic Bacteremia With Positive L. Reuteri Identification
Description: The presence of symptomatic bacteremia with positive L. reuteri identification was assessed and none of the participants in either group showed any clinical features of suspected bacteremia in this study.
Time Frame: Approximately 98 days
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | SB-121 | Placebo
Number analyzed (Participants) | 15 | 15
Participants | 0 | 0

4. Secondary Outcome: Mean Percent Change From Baseline in Biomarkers: Tumor Necrosis Factor-α
Description: Mean (standard deviation) percent changes from baseline in tumor necrosis factor-α
Time Frame: Day -28 to Day 0, Period 1: Day 28; Period 2: Days 1 (pre-dose) and 28 (period = 28 days and 14 days wash-out)
Population: Safety Population.
  To be noted changes at crossover in N:
  Treatment Period 1 - SB-121 (N=7) and Placebo (N=8) Treatment Period 2 - SB-121 (N=8) and Placebo (N=7)
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | SB-121 | Placebo
Number analyzed (Participants) | 15 | 15
percentage
  changes from baseline to Treatment Period 1 (Day 28): number analyzed (Participants) | 7 | 8
  changes from baseline to Treatment Period 1 (Day 28) | 37.98 (57.70) | 0.27 (23.23)
  changes from baseline to Treatment Period 2 (Day 28/end of treatment): number analyzed (Participants) | 8 | 7
  changes from baseline to Treatment Period 2 (Day 28/end of treatment) | -1.11 (16.51) | 8.77 (50.41)

5. Secondary Outcome: Mean Percent Change From Baseline in Biomarkers: Serum High-sensitivity C-reactive Protein (Hs-CRP)
Description: Mean (standard deviation) percent change from baseline in serum high-sensitivity C-reactive protein (hs-CRP)
Time Frame: Day -28 to Day 0, Period 1: Day 28; Period 2: Days 1 (pre-dose) and 28 (period = 28 days and 14 days wash-out)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | SB-121 | Placebo
Number analyzed (Participants) | 15 | 15
percent
  changes from baseline to Treatment Period 1 (Day 28): number analyzed (Participants) | 7 | 7
  changes from baseline to Treatment Period 1 (Day 28) | 173.38 (306.88) | 45.70 (118.29)
  changes from baseline to Treatment Period 2 (Day 28/end of treatment): number analyzed (Participants) | 8 | 7
  changes from baseline to Treatment Period 2 (Day 28/end of treatment) | -13.91 (40.56) | -33.13 (30.52)

6. Secondary Outcome: Mean Percent Change From Baseline in Biomarkers: Stool Biomarkers, Fecal Calprotectin
Description: Mean (standard deviation) percent change from baseline in stool biomarkers, fecal calprotectin.
  The number of participants with data available are presented.
Time Frame: Period 1: Days 1 (pre-dose), 28 and 35; Period 2: Days 28 and 35 (period = 28 days and 14 days wash-out)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | SB-121 | Placebo
Number analyzed (Participants) | 15 | 15
percent
  changes from baseline to Treatment Period 1 (Day 28): number analyzed (Participants) | 4 | 5
  changes from baseline to Treatment Period 1 (Day 28) | 76.1 (99.79) | 2.7 (67.29)
  changes from baseline Treatment Period 2 (Day 28/end of treatment): number analyzed (Participants) | 4 | 4
  changes from baseline Treatment Period 2 (Day 28/end of treatment) | -39.9 (25.21) | -26.1 (21.78)
  changes from baseline Treatment Period 2 (Day 42/poststudy washout): number analyzed (Participants) | 5 | 4
  changes from baseline Treatment Period 2 (Day 42/poststudy washout) | -4.2 (35.56) | -14.0 (25.43)

7. Secondary Outcome: Mean Percent Change From Baseline in Biomarkers: Stool Biomarkers, Fecal Lactoferrin
Description: Mean (standard deviation) percent change from baseline in stool biomarkers, fecal lactoferrin.
  The number of participants with data available are presented.
Time Frame: Period 1: Days 1 (pre-dose), 28 and 35; Period 2: Days 28 and 35 (period = 28 days and 14 days wash-out)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | SB-121 | Placebo
Number analyzed (Participants) | 15 | 15
percent
  change from baseline to Treatment Period 1 (Day 28): number analyzed (Participants) | 3 | 5
  change from baseline to Treatment Period 1 (Day 28) | NA (NA) — NA = 0.0. The reason these values are "0" is a combination of: 1) There were a lot stool samples missing so most do not have both pre and post sample values, and 2) values below the LLQ parameter are reported as 1.000 which was the case for most samples. | 49.40 (110.46)
  change from baseline to Treatment Period 2 (Day 28/end of treatment): number analyzed (Participants) | 4 | 3
  change from baseline to Treatment Period 2 (Day 28/end of treatment) | 12.33 (36.63) | -42.90 (35.75)
  change from baseline to Treatment Period 2 (Day 42/poststudy washout): number analyzed (Participants) | 5 | 3
  change from baseline to Treatment Period 2 (Day 42/poststudy washout) | 47.08 (105.57) | -40.97 (34.52)

8. Secondary Outcome: Mean Percent Change From Baseline in Biomarkers: Plasma Oxytocin
Description: The mean (standard deviation) percent changes from baseline in plasma oxytocin.
Time Frame: Day -28 to Day 0, Period 1: Day 28; Period 2: Days 1 and 28 (period = 28 days and 14 days wash-out)
Population: Safety Population
  To be noted changes at crossover in N:
  Treatment Period 1 - SB-121 (N=7) and Placebo (N=8) Treatment Period 2 - SB-121 (N=8) and Placebo (N=7)
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | SB-121 | Placebo
Number analyzed (Participants) | 15 | 15
percent
  change from baseline to Treatment Period 1 (Day 28): number analyzed (Participants) | 7 | 7
  change from baseline to Treatment Period 1 (Day 28) | 178.83 (167.54) | 61.69 (95.04)
  change from baseline to Treatment Period 2 (Day 28/end of treatment): number analyzed (Participants) | 7 | 6
  change from baseline to Treatment Period 2 (Day 28/end of treatment) | 44.43 (118.64) | -18.53 (26.92)

9. Secondary Outcome: Mean Percent Change From Baseline in Biomarkers: Plasma Vasopressin
Description: Mean (standard deviation) percent changes from baseline in plasma vasopressin levels
Time Frame: Day -28 to Day 0, Period 1: Day 28; Period 2: Days 1 (pre-dose) and 28 (period = 28 days and 14 days wash-out)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | SB-121 | Placebo
Number analyzed (Participants) | 15 | 15
percent
  change from baseline to Treatment Period 1 (Day 28): number analyzed (Participants) | 7 | 7
  change from baseline to Treatment Period 1 (Day 28) | 55.98 (115.43) | 16.53 (41.70)
  change from baseline to Treatment Period 2 (Day 28/end of treatment): number analyzed (Participants) | 7 | 6
  change from baseline to Treatment Period 2 (Day 28/end of treatment) | -10.14 (27.80) | 21.36 (72.46)

ADVERSE EVENTS:
Time Frame: Any time after informed consent was obtained until 14 days after study treatment, approximately 14 weeks (112 days)
Description: The study team recorded all adverse events (AEs) with start dates occurring any time after informed consent was obtained until 14 days after study treatment. At each study visit, the study team asked about the occurrence of AEs since the last visit whether in the clinic or on the phone.
Groups:
- SB-121: Includes all participants who received SB-121, whether in Treatment Period 1 or 2.
- Placebo: Includes all participants who received placebo, whether in Treatment Period 1 or 2.
Arm/Group | SB-121 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 7/15 | 9/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB-121 (N=15) | Placebo (N=15)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 3 (5)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 (2)
Fatigue (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Sinusitis (Infections and infestations) | 2 | 0
COVID-19 (Infections and infestations) | 0 | 1
Tinea infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Bilirubinuria (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT04944901/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT04944901/SAP_001.pdf